CLINICAL TRIAL: NCT03578289
Title: Efficacy and Feasibility of a Tele-mental Health Intervention to Support Parents Caring for a Technology-dependent Child at Home
Brief Title: A Tele-mental Health Intervention to Support Parents Caring for a Technology-dependent Child at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Yudy Muneton-Castano, Clinical Social Worker, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00023319
Record Dates: First submitted 2016-11-08; First posted 2018-07-06 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Mental Fatigue
Keywords: Parents of children with disabilities; emotional functioning
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (telemental health_ (Experimental): The experimental group will received cognitive behavioral therapy (CBT) via TMH for 8 sessions.
  Interventions: Behavioral: Telemental Health - CBT
- Waiting Control Group (usual care) (Experimental): Participants randomly assigned to the control group will receive routine care for three months followed by the 8-week CBT intervention
  Interventions: Behavioral: Telemental Health - CBT

INTERVENTIONS:
Behavioral: Telemental Health - CBT — The experimental group will received cognitive behavioral therapy (CBT) via TMH for 8 sessions.

SUMMARY:
The need for assisted-technology at home reflects some of the most serious health-related conditions faced by children with physical and developmental disabilities. 'Technology-dependent' is often used in the literature to describe children "who need both a medical device to compensate for the loss of a vital body function and substantial and ongoing nursing care to avert death or further disability". Parenting a child is stressful and challenging, and even under ideal circumstances the care of a child with complex needs requires greater than normal parenting skills. Studies have showed that parents of children whose illness require assisted-technology experience significant emotional stress, potential gaps in social support, and social isolation leading to lower quality of life, unhealthy family functioning, and negative psychological consequences.

This study intends to assess the feasibility and efficacy of a tele-psychotherapy (Tele-P) intervention as a way to promote the emotional functioning of parents and to help increase the quality of life of children that are technology-dependent in the Greater Boston Area. It is hypothesized that parents who adhere to psychotherapy sessions via videoconferencing (Tele-P) will demonstrate significant reductions in symptoms of depression, anxiety and social isolation. Children of parents in the (Tele-P) condition will show significantly greater improvements in their quality of life including their physical health, mental health, family life, free time, and general life enjoyment.

A randomized controlled trial is proposed in order to evaluate the feasibility and efficacy of a tele-psychotherapy intervention for parents of technology-dependent children at the Critical Care, Anesthesia and Perioperative Extension (CAPE) program in Boston Children's Hospital.

This study will serve as model for social workers to perform an intervention for parent's raising technology-dependent children. This study proposes that tele-psychotherapy be a means of advocating for this underserved population.

DETAILED DESCRIPTION:
Efficacy and Feasibility of a tele-psychotherapy intervention to support parents caring for a technology-dependent child at home.

Caring for a technology-dependent child at home is a challenging experience for parents. Global family functioning, lifestyles changes and vocational decisions are affected. Parents of children whose chronic illness require assisted-technology experience significant emotional stress, potential gaps in social support, and social isolation leading to lower quality of life, unhealthy family functioning, and negative psychological consequences.

This study intends to evaluate a tele-psychotherapy (Tele-P) intervention as a way to promote the emotional functioning of parents and secondarily increase the quality of life of children that are home technology-dependent in the Greater Boston Area. The sample will consist of parents of children that are technology-dependent in the Critical Care, Anesthesia and Perioperative Extension (CAPE) Program at Boston Children's Hospital.

Specific Aim 1) To assess the feasibility of delivering a cognitive behavioral Tele-P intervention for parents of children that are technology-dependent in the Critical Care, Anesthesia and Perioperative Extension (CAPE) Program at Boston Children's Hospital.

Hypothesis 1: Parents and therapist will adhere to 8 psychotherapy sessions via videoconferencing.

Hypothesis 2: Cost analysis evaluation will validate the feasibility of the intervention vs. usual care (UC) and standard face-to-face therapy sessions.

Specific Aim 2) To evaluate the efficacy of a Tele-P intervention relative to UC in management of mental health conditions amongst parents of children with chronic respiratory failure.

Hypothesis 1: Relative to parents assigned to the UC condition, those in the (Tele-P) condition will: a) demonstrate significant reductions in symptoms of depression, b) significant reductions in symptoms of anxiety and c) significantly less social isolation.

Hypothesis 2: Improvement in mental health symptoms will be sustained for the duration of therapy.

Specific Aim 3) To assess whether a Tele-P intervention increases the quality of life of children in the Critical Care, Anesthesia and Perioperative Extension (CAPE) Program at Boston Children's Hospital.

Hypothesis 1: Children of parents participating in Tele-P will show significantly greater improvements in their quality of life relative to their UC counterparts on outcomes of a) physical health, b) mental health (happiness, wellbeing), c) family life, d) free time, and e) general life enjoyment.

Background and Significance

'Technology-dependent' is often used in the literature to describe children "who need both a medical device to compensate for the loss of a vital body function and substantial and ongoing nursing care to avert death or further disability". Approximately 1.2 million children and adolescents in the United States require durable medical equipment to survive. In the early 1990's, surveys estimated that over 2,200 children in Massachusetts were dependent upon some degree of assisted medical technology. The number of ventilator-dependent children in the Boston community had since increased threefold, representing increased survival of low birth weight infants and those with chronic life-limiting illnesses. Recent studies have shown that technology-dependent children comprise 20% of all pediatric patients discharged from the hospital to home, yet they account for 61% of all healthcare resources used by children. While advances in medical care have brought children with chronic health conditions life-saving and sustaining advances, healthcare systems are inadequately structured to meet their ongoing comprehensive needs. Most of these children are cared for at home by parents and have substantial functional limitations including: self-care, self-direction, capacity for independent living and economic self-sufficiency.

The need for assisted technology at home reflects some of the most serious health-related conditions faced by children with physical and developmental disabilities and their parents. Parenting a child is stressful and challenging, and even under ideal circumstances the care of a child with complex needs requires greater than normal parenting skills. Parents assume an altered parental role, serving as parent, care coordinator, respiratory therapist, nurse, and any other function that is required for 24 hour a day care. The cost of medical care, prescriptions, and durable medical equipment effects families independent of their employment and insurance states. This causes an even greater burden on these already financially, emotionally, and physically stressed parents. Prospects of independence, self-care, self-direction with growth are not viable for some of these children, contributing to an indeterminate need for parental effort. Cumulative toll impacts all members of the family and may also impact medical outcomes

The investigators previous work showed that the parents of children whose chronic illness require assisted-technology experience significant emotional stress, potential gaps in social support, and social isolation leading to lower quality of life, unhealthy family functioning, and negative psychological consequences. Approximately 36-45% of mothers caring for technology dependent children have an escalated risk for clinical depression. Sleep deprivation due to anxiety about a child's condition, false monitor alarms, and the need to remain vigilant over the child during the night is a common theme for parents of technology dependent children. Data suggests sleep disruption places family caregivers at risk for poor health and related outcomes that may impair their daytime function and long term capacity for caregiving. Raising a technology-dependent child significantly impacts family functioning and hence the quality of life outcomes for the family. Depression and anxiety in parents negatively affects the quality of care a parent can provide their child. Young children exposed to depressed parents run a risk for delay in language, personal social gross motor, and fine motor development. Increase perceived parental burden and consequent family impact may result in negative implications on their own and their children's health related quality of life. Support for parents is crucial not only for the course of the disease of the child but also for the parents' health.

In the Greater Boston area there are limited specialized mental health resources and it is increasingly difficult for parents of children that are technology-dependent to obtain appropriate mental health treatment. Social workers currently have few evidence-based inventions tested on families with chronically ill children. Immediate action is necessary to provide resources to parents to help them feel motivated, confident and capable of caring for a child. These children are extremely vulnerable and it is imperative to their quality of life that their parents are capable of providing appropriate care. This proposal intends to address this gap in parental care through Tele-P, a unique therapy via video conference, to help parents cope with these daily stressors. As feelings of depression, anxiety and social isolation decrease, parents should feel more confident and capable of caring for their child. Technology dependent children fully rely on their caregivers in order to not only improve their health but to survive. As Tele-P improves the mental health of the parent, the child's care and quality of life will also greatly improve.

Tele-P can be successfully used in several therapeutic formats, has similar outcomes as face to face treatment, and is considered satisfactory by most patients and therapist. There are proven to be a number of benefits to home based tele-mental health including better adherence to appointments, overcoming social isolation, access to contextual information such as the patient's home situation, improved patient and practitioner safety and removal of fears and stigma attached to attending a mental health clinic. Providing therapy through videoconferencing relieves the parents from the stress of traveling with their technology dependent children, which often requires time, resources, (such as an ambulance) and money. For some technology-dependent children it is also dangerous for them to travel due to their severe diagnosis. Tele-P allows for the parents to be at home with their child, but at the same time be part of a social interaction. Studies have shown that "facing a high burden of care but still being able to have sufficient social and familial contacts seems to be somewhat protective regarding the mental health of these parents, pointing even stronger towards the importance of social integration". Tele-P is a unique acceptable and sustainable approach to address the gap in access to services for underserved populations. Feasibility remains a question. The investigators experience with survey completion in this population suggests that time and care demands may be a limiting factor. Given the option of electronic paper survey in a previous study, the majority completed the latter despite computer access. Paper was easier to interrupt and resume if the child's care was needed.

There is an urgent need for support of parents with technology-dependent children. Although researchers have identified a plethora of risks, stressors, and needs of the families with chronically ill child, there is a scarcity of evidence based interventions that address the mental health needs of parents or caregivers of children with developmental disabilities. Providing Tele-P is a well-suited approach for these parents and caregivers, who may be overwhelmed by their children's situation, anticipating future challenges and reliving past traumas. The results of the Tele-P sessions could also be a valuable tool to guide intervention with policies, resources and services that may improve family quality of life and outcomes for families who are raising children with developmental disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child cared for in the CAPE Program
* 18 years of age or older
* Lack of active mental health counseling
* English or Spanish speaking

Exclusion Criteria:

* History of psychosis in the past six months
* Receipt of any mental health treatment within the 3 months prior to study enrollment
* Future appointment with a mental health provider within the next two months and evidence of suicidal thoughts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Number of participants in the intervention | 12 Months
  Number of participants who complete the intervention

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information Systems (PROMIS) Global Scale | 12 Months
  Change in PROMIS Global Scale from baseline to post intervention. This is a 10 item scale. Higher scores will correspond to better feasibility and acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided